CLINICAL TRIAL: NCT00996476
Title: A Phase II, Randomized, Open-label Study in Japan to Investigate the Efficacy, Safety and Pharmacokinetics of TMC435 as Part of a Treatment Regimen Including Peginterferon Alfa-2a and Ribavirin in Treatment naïve, Genotype 1, Chronic Hepatitis C Subjects
Brief Title: A Study to Assess the Effectiveness, Safety, and Pharmacokinetics of TMC435 in Combination With Peginterferon Alfa-2a and Ribavirin in Hepatitis-C Infected Patients
Acronym: DRAGON
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR016402; TMC435-TiDP16-C215 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Results first posted 2014-04-17 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-03

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis C; Hepatitis C virus; Interferon Alfa-2a; Ribavirin; Viral RNA
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — Simeprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- TMC12/PR24 50 mg (Experimental): Participants received TMC435 50 mg once daily with PegIFNa-2a and ribavirin (PR) for 12 weeks followed by PR until Week 24 Participants who achieved plasma hepatitis C virus (HCV) ribonucleic acid (RNA) levels <1.4 log10 IU/mL at Week 4 and had undetectable plasma HCV RNA at Weeks 12, 16 and 20, discontinued all study treatment (TMC435 and PR) at Week 24. All other participants continued PR until Week 48.
  Interventions: Drug: TMC435; Drug: PegIFNα-2a; Drug: RBV
- TMC12/PR24 100 mg (Experimental): Participants received TMC435 100 mg once daily plus PegIFNa-2a and ribavirin (PR) for 12 weeks followed by PR until Week 24. Participants who achieved plasma hepatitis C virus (HCV) ribonucleic acid (RNA) levels <1.4 log10 IU/mL at Week 4 and had undetectable plasma HCV RNA at Weeks 12, 16 and 20, discontinued all study treatment (TMC435 and PR) at Week 24. All other participants continued PR until Week 48.
  Interventions: Drug: TMC435; Drug: PegIFNα-2a; Drug: RBV
- TMC24/PR24 50 mg (Experimental): Participants received TMC435 50 mg once daily plus PegIFNa-2a and ribavirin (PR) for 24 weeks. Participants who achieved plasma hepatitis C virus (HCV) ribonucleic acid (RNA) levels <1.4 log10 IU/mL at Week 4 and had undetectable plasma HCV RNA at Weeks 12, 16 and 20, discontinued all study treatment (TMC435, PR) at Week 24. All other participants continued PR until Week 48.
  Interventions: Drug: TMC435; Drug: PegIFNα-2a; Drug: RBV
- TMC24/PR24 100 mg (Experimental): Participants received TMC435 100 mg once daily plus PegIFNa-2a and ribavirin (PR) for 24 weeks. Participants who achieved plasma hepatitis C virus (HCV) ribonucleic acid (RNA) levels <1.4 log10 IU/mL at Week 4 and had undetectable plasma HCV RNA at Weeks 12, 16 and 20, discontinued all study treatment (TMC435 and PR) at Week 24. All other participants continued PR until Week 48.
  Interventions: Drug: TMC435; Drug: PegIFNα-2a; Drug: RBV
- PR48 Control (Experimental): Participants received PegIFNa-2a and ribavirin (PR) for 48 weeks (PR48 control group)
  Interventions: Drug: TMC435; Drug: PegIFNα-2a; Drug: RBV

INTERVENTIONS:
Drug: TMC435 — One 50 or 100-mg capsule orally (by mouth), once daily for 12 or 24 weeks
Drug: PegIFNα-2a — One subcutaneous injection of PegIFNα-2a 180 μg once weekly for 12, 24, or 48 weeks.
Drug: RBV — 300, 400, or 500-mg tablets orally twice daily for 12, 24, or 48 weeks.

SUMMARY:
The purpose of this study is to evaluate effectiveness, safety and pharmacokinetics (Explores what the body does to the medication) of TMC435350 in combination with Peginterferon Alfa-2a and Ribavirin in genotype 1 hepatitis C virus infected Japanese participants who have never received treatment for their hepatitis C infection.

DETAILED DESCRIPTION:
This is a Phase 2, randomized (The study medication is assigned by chance.), 5-arm, open label (All people know the identity of the intervention.), multicentre (study conducted at multiple sites) study. Approximately, 84 participants will be randomized to 5 different arms in a 2:2:1:1:1 ratio. In treatment arms 1 and 2, participants will receive 12 weeks of triple therapy (use of 3 medications) with TMC435 50 or 100 mg once daily plus Peginterferon Alfa-2a and Ribavirin followed by 12 weeks of treatment with Peginterferon Alfa-2a and Ribavirin. In treatment arms 3 and 4, participants will receive 24 weeks of triple therapy with TMC435 50 or 100 mg once daily plus Peginterferon Alfa-2a and Ribavirin. In treatment arm 5 (control group), participants will receive Peginterferon Alfa-2a and Ribavirin for 48 weeks. This study will consist a screening phase of upto 6 weeks, treatment phase of upto 48 weeks and a post treatment follow-up period of 24 weeks. Safety evaluations will include assessment of adverse events, clinical laboratory tests, vital signs, and cardiovascular safety.

ELIGIBILITY:
Inclusion Criteria:

* Participants with documented chronic hepatitis C infection as evidenced by presence of HCV antibody at least 6 months (180 days) prior to the informed consent. - Participants with genotype 1 HCV infection. - Participants with plasma HCV RNA level of ≥ 5.0 log10 IU/mL at screening.

Exclusion Criteria:

* Participants diagnosed with hepatic cirrhosis or hepatic failure. - Participants with any other liver disease than hepatitis C. - Participants with infection/co-infection with non-genotype 1 HCV.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2009-07; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K. Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (19):
- Japan (19):
  - Amagasaki
  - Hiroshima
  - Kagoshima
  - Kawasaki
  - Kitakyushu
  - Kurume
  - Kyoto
  - Matsumoto
  - Musashino
  - Nishinomiya
  - Ohmura
  - Osaka
  - Ōsaka-sayama
  - Sakai
  - Sapporo
  - Suita
  - Tokyo
  - Touon
  - Yokohama

REFERENCES:
- [Derived] Hayashi N, Seto C, Kato M, Komada Y, Goto S. Once-daily simeprevir (TMC435) with peginterferon/ribavirin for treatment-naive hepatitis C genotype 1-infected patients in Japan: the DRAGON study. J Gastroenterol. 2014 Jan;49(1):138-47. doi: 10.1007/s00535-013-0875-1. Epub 2013 Sep 5. PMID 24005956

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between 6 July 2009 and 1 April 2011 and recruited participants with chronic Hepatitis C Virus (HCV) infection from 25 study centers in Japan. A total of 93 participants were randomized, 92 treated, and 85 completed the study (1 participant in the TMC12/PR24 100 mg arm withdrew consent and did not receive study treatment).
Pre-assignment Details: Treatment-naïve HCV-infected participants were randomized to 1 of 5 treatment arms and received 12 weeks of TMC435 50 or 100 mg once daily with PegIFNα-2a and ribavirin (PR) followed by 12 weeks of PR (Arm 1 and 2); 24 weeks of TMC435 50 or 100 mg once daily with PR (Arms 3 and 4); and, PR for 48 weeks (Arm 5).
Period: Overall Study
Arm/Group | TMC12/PR24 50 mg | TMC12/PR24 100 mg | TMC24/PR24 50 mg | TMC24/PR24 100 mg | PR48 Control
Started | 27 | 26 | 13 | 13 | 13
Completed | 26 | 23 | 12 | 13 | 11
Not Completed | 1 | 3 | 1 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 2 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TMC12/PR24 50 mg | TMC12/PR24 100 mg | TMC24/PR24 50 mg | TMC24/PR24 100 mg | PR48 Control | Total
Number analyzed (Participants) | 27 | 26 | 13 | 13 | 13 | 92
Age, Continuous [Median (Full Range); unit: years] | 53 [31 to 67] | 56 [22 to 69] | 48 [34 to 67] | 54 [28 to 68] | 54 [20 to 66] | 54 [20 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 7 | 5 | 6 | 49
  Male | 12 | 10 | 6 | 8 | 7 | 43

OUTCOME MEASURES:

1. Primary Outcome: Change in Plasma Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Levels From Baseline to Week 4
Description: The table below shows the least-squares (LS) mean change and 95% confidence intervals (CI) change from baseline at Week 4 in HCV RNA levels for participants in the 2 TMC435 50 mg treatment groups combined (TMC12/PR24 50 mg and TMC24/PR24 50 mg) and for participants in the 2 TMC435 100 mg treatment groups combined (TMC12/PR24 100 mg and TMC24/PR24 100 mg). The statistical analyses show the difference in LS mean change from baseline from the PR48 control group and the 95% CI for each dose group (ie, each TMC435 dose group minus PR48 control). NOTE: All outcome measures reported in this study are "Exploratory;" not "Primary" as indicated (refer to Limits and Caveats).
Time Frame: Day 1 (Baseline) and Week 4
Population: The efficacy analyses were based on the per protocol set (PPS) of participants and consisted of a subset of participants in the full analysis set (FAS) which had no major protocol violations suspected to influence efficacy assessment and had data available at the time point(s) analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: log10 IU/mL
Groups:
- TMC435 50 mg: Participants who received TMC435 50 mg in Treatment Groups TMC12/PR24 50 mg and TMC24/PR24 50 mg
- TMC435 100 mg: Participants who received TMC435 100 mg in Treatment Groups TMC12/PR24 100 mg and TMC24/PR24 100 mg
- PR48 Control: Participants received PegIFNα-2a and ribavirin (PR) for 48 weeks (PR48 control group)
Arm/Group | TMC435 50 mg | TMC435 100 mg | PR48 Control
Number analyzed (Participants) | 39 | 37 | 11
log10 IU/mL | -5.23 (0.55) [-5.43 to -5.02] | -5.24 (0.47) [-5.45 to -5.03] | -2.83 (1.93) [-3.21 to -2.45]
Statistical Analysis 1: Comparison: TMC435 50 mg vs PR48 Control; Difference in least square (LS) mean change from baseline from the PR48 control group; Test type: Superiority or Other; ANCOVA; LS means difference = -2.40, 95% CI 2-sided [-2.83 to -1.97] — TMC435 50 mg minus PR48 control
Statistical Analysis 2: Comparison: TMC435 100 mg vs PR48 Control; Difference in least square (LS) mean change from baseline from the PR48 control group; Test type: Superiority or Other; ANCOVA; LS Means difference = -2.41, 95% CI 2-sided [-2.85 to -1.98] — TMC435 100 mg minus PR48 control

2. Primary Outcome: The Percentage of Participants With Undetectable Plasma Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Levels During the Study
Description: The table below shows the percentage of participants in each treatment group with undetectable plasma HCV RNA levels at Weeks 4, 12, 24, 48, and end of treatment (EOT, up to Week 24 or 48). The number of participants analyzed is listed at each time point in order of the treatment groups from left to right in the table (ie, Week x, n=x, x, x, x, and x) if different from the "Number of Participants Analyzed."NOTE: All outcome measures reported in this study are "Exploratory;" not "Primary" as indicated (refer to Limits and Caveats).
Time Frame: Weeks 4, 12, 24 or 48, and EOT (up to Week 24 or 48)
Population: Efficacy analyses were based on the per protocol set (PPS) of participants and consisted of a subset of participants in the full analysis set (FAS) which had no major protocol violations suspected to influence efficacy assessment and had data available at the time point(s) analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | TMC12/PR24 50 mg | TMC12/PR24 100 mg | TMC24/PR24 50 mg | TMC24/PR24 100 mg | PR48 Control
Number analyzed (Participants) | 27 | 24 | 13 | 13 | 11
Percentage of participants
  Week 4 (n=27, 24, 12, 13, and 11) | 85.2 | 100.0 | 83.3 | 92.3 | 9.1
  Week 12 (n=27, 22, 12, 13, and 11) | 100.00 | 100.0 | 100.0 | 100.0 | 54.45
  Week 24 (n=26, 21, 11, 13, and 11) | 96.2 | 100.0 | 100.0 | 100.0 | 81.8
  Week 48 (n=25, 20, 12, 13, and 10) | 80.0 | 95.0 | 83.3 | 92.3 | 90.0
  EOT (up to Week 24 or 48) | 96.3 | 100.0 | 92.3 | 100.0 | 90.9

3. Primary Outcome: The Percentage of Participants With a Decrease of Greater Than or Equal to 2 log10 IU/mL From Baseline in Plasma Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Through the Post-treatment Follow-up Period
Description: The table below shows the percentage of participants in each treatment group with a decrease of greater than (>) or equal (=) to 2 log10 IU/mL from baseline in plasma HCV RNA levels at time points during the treatment period and post treatment follow-up period. The number of participants analyzed is listed at each time point in order of the treatment groups from left to right in the table (ie, Week x, n=x, x, x, x, and x) if different from the "Number of Participants Analyzed." NOTE: All outcome measures reported in this study are "Exploratory;" not "Primary" as indicated (refer to Limits and Caveats).
Time Frame: Days 1 (4 hr), 1 (8 hr), 3, Weeks 1, 2, 3, 4, 6, 8, 12, 16, 20, 24,28, 36, 42, 48, 52, 60, 72, and EOT (up to Week 24 or 48)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | TMC12/PR24 50 mg | TMC12/PR24 100 mg | TMC24/PR24 50 mg | TMC24/PR24 100 mg | PR48 Control
Number analyzed (Participants) | 27 | 24 | 13 | 13 | 11
Percentage of participants
  Day 1 (4hr) | NA — no participants were analyzed for this time point | NA — no participants were analyzed for this time point | NA — no participants were analyzed for this time point | NA — no participants were analyzed for this time point | NA — no participants were analyzed for this time point
  Day 1 (8hr) | NA — no participants were analyzed for this time point | NA — no participants were analyzed for this time point | NA — no participants were analyzed for this time point | NA — no participants were analyzed for this time point | NA — no participants were analyzed for this time point
  Day 3 | 100.0 | 100.0 | 92.3 | 92.3 | 18.2
  Week 1 | 100.0 | 100.0 | 100.0 | 100.0 | 27.3
  Week 2 (n=27, 24, 12, 13, and 11) | 100.0 | 100.0 | 100.0 | 100.0 | 54.5
  Week 3 (n=27, 24, 12, 13, and 11) | 100.0 | 100.0 | 100.0 | 100.0 | 54.5
  Week 4 (n=27, 24, 12, 13, and 11) | 100.0 | 100.0 | 100.0 | 100.0 | 54.5
  Week 6 (n=27, 23, 12, 13, and 11) | 100.0 | 100.0 | 100.0 | 100.0 | 72.7
  Week 8 (n=27, 22, 12, 13, and 11) | 100.0 | 100.0 | 100.0 | 100.0 | 81.8
  Week 12 (n=27, 22, 12, 13, and 11) | 100.0 | 100.0 | 100.0 | 100.0 | 81.8
  Week 16 (n=26, 22, 12, 13, and 11) | 100.0 | 95.5 | 100.0 | 100.0 | 90.9
  Week 20 (n=26, 22, 12, 13, and 11) | 100.0 | 95.5 | 100.0 | 100.0 | 90.9
  Week 24 (n=26, 21, 11, 13, and 11) | 96.2 | 100.0 | 100.0 | 100.0 | 90.9
  Week 28 (n=26, 21, 11, 13, and 11) | 92.3 | 95.2 | 100.0 | 100.0 | 90.9
  Week 36 (n=26, 21, 12, 13, and 11) | 88.5 | 95.2 | 91.7 | 92.3 | 90.9
  Week 42 (0, 0, 0, 0, and 10) | NA — no participants were analyzed for this time point | NA — no participants were analyzed for this time point | NA — no participants were analyzed for this time point | NA — no participants were analyzed for this time point | 90.0
  Week 48 (25, 20, 12, 13, and 10) | 80.0 | 95.0 | 91.7 | 92.3 | 100.0
  EOT (n=27, 24, 13, 13, and 11) | 96.3 | 100.0 | 100.0 | 100.0 | 90.9
  Week 52 ((n=0, 0, 0, 0, and 9) | NA — no participants were analyzed for this time point | NA — no participants were analyzed for this time point | NA — no participants were analyzed for this time point | NA — no participants were analyzed for this time point | 88.9
  Week 60 (0, 0, 0, 0, and 9) | NA — no participants were analyzed for this time point | NA — no participants were analyzed for this time point | NA — no participants were analyzed for this time point | NA — no participants were analyzed for this time point | 55.6
  Week 72 (0, 0, 0, 0, and 8) | NA — no participants were analyzed for this time point | NA — no participants were analyzed for this time point | NA — no participants were analyzed for this time point | NA — no participants were analyzed for this time point | 62.5

4. Primary Outcome: The Percentage of Participants With Plasma Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Levels Undetectable or Below the Limit of Quantification (<1.2 log10 IU/mL Detectable) During Treatment and During Post Treatment Follow-up
Description: The table below shows the percentage of participants in each treatment group with plasma HCV RNA levels undetectable or below the limit of quantification (<1.2 log10 IU/mL detectable ) at time points during treatment and post treatment follow-up.The number of participants analyzed is listed at each time point in order of the treatment groups from left to right in the table (ie, Week x, n=x, x, x, x, and x) if different from the "Number of Participants Analyzed." NOTE: All outcome measures reported in this study are "Exploratory;" not "Primary" as indicated (refer to Limits and Caveats).
Time Frame: Week 4, 12, 24, 36, 48, EOT (up to Week 24 or 48), and Week 60 and 72
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | TMC12/PR24 50 mg | TMC12/PR24 100 mg | TMC24/PR24 50 mg | TMC24/PR24 100 mg | PR48 Control
Number analyzed (Participants) | 27 | 24 | 13 | 13 | 11
Percentage of participants
  Week 4 (n=27, 24,12,13, and 11) | 100.0 | 100.0 | 100.0 | 100.0 | 18.2
  Week 12 (n=27, 22, 12, 13, and 7) | 100.0 | 100.0 | 100.0 | 100.0 | 81.8
  Week 24 (n=26, 21, 11, 13, and 11) | 96.2 | 100.0 | 100.0 | 100.0 | 81.8
  Week 36 (n=26, 21, 11, 12, and 11) | 88.5 | 90.5 | 91.7 | 92.3 | 90.9
  Week 48 (n=25, 20, 12, 13, and 10) | 80.0 | 95.0 | 83.3 | 92.3 | 90.0
  EOT (up to Week 24 or 48) | 96.3 | 100.0 | 100.0 | 100.0 | 90.9
  Week 60 (n=0,0,0,0, and 9) | NA — no participants were analyzed for this time point | NA — no participants were analyzed for this time point | NA — no participants were analyzed for this time point | NA — no participants were analyzed for this time point | 55.6
  Week 72 (n=0,0,0,0, and 8) | NA — no participants were analyzed for this time point | NA — no participants were analyzed for this time point | NA — no participants were analyzed for this time point | NA — no participants were analyzed for this time point | 62.5

5. Primary Outcome: The Number of Participants With Viral Breakthrough
Description: The table below shows the number of participants in each treatment group who experienced viral breakthrough during the 48 week treatment period with at least one study medication (TMC435 or PegIFNα-2a and ribavirin). Viral breakthrough is defined as a confirmed increase of greater than (>) 1 log10 IU/mL in plasma hepatitis C virus (HCV) ribonucleic acid (RNA) level from the lowest level reached or a confirmed value of plasma HCV RNA of > 2.0 log10 IU/mL in participants whose plasma HCV RNA level had previously been reported below 1.2 log10 IU/mL detectable or undetectable during the treatment period. The number of participants analyzed is listed at each time point in order of the treatment groups from left to right in the table (ie, Week x, n=x, x, x, x, and x) if different from the "Number of Participants Analyzed." NOTE: All outcome measures reported in this study are "Exploratory;" not "Primary" as indicated (refer to Limits and Caveats).
Time Frame: Up to EOT (up to Week 24 or 48)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | TMC12/PR24 50 mg | TMC12/PR24 100 mg | TMC24/PR24 50 mg | TMC24/PR24 100 mg | PR48 Control
Number analyzed (Participants) | 27 | 24 | 13 | 13 | 11
Participants | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: The Percentage of Participants With Viral Relapse
Description: The table below shows the percentage of participants in each treatment group who experienced viral relapse within 12 weeks (ie, at Week 36 or 60) after actual end of treatment (EOT) (up to Week 24 or 48). Viral relapse was defined as confirmed detectable plasma hepatitis C virus (HCV) ribonucleic acid (RNA) levels during the post treatment follow-up period at Weeks 36 or 60 in participants with undetectable plasma HCV RNA at EOT. The statistical analysis shows the difference in treatments (ie, each TMC435 group minus PR48 control) in viral relapse. NOTE: All outcome measures reported in this study are "Exploratory;" not "Primary" as indicated (refer to Limits and Caveats).
Time Frame: Week 36 or 60
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | TMC12/PR24 50 mg | TMC12/PR24 100 mg | TMC24/PR24 50 mg | TMC24/PR24 100 mg | PR48 Control
Number analyzed (Participants) | 26 | 24 | 12 | 13 | 10
Participants | 15.4 | 12.5 | 16.7 | 7.7 | 40.0
Statistical Analysis 1: Comparison: TMC12/PR24 50 mg vs PR48 Control; The difference in the percentage of participants between The TMC12/PR24 50 mg treatment group and the PR48 control group; Test type: Superiority or Other; Difference in percentage of participants = -24.6, 95% CI 2-sided [-58.3 to 11.8] — PR48 control minus TMC12/PR24
Statistical Analysis 2: Comparison: TMC12/PR24 100 mg vs PR48 Control; The difference in the percentage of participants between The TMC12/PR24 100 mg treatment group and the PR48 control group; Test type: Superiority or Other; Difference in percentage of participants = -27.5, 95% CI 2-sided [-61.1 to 9.8] — PR48 control minus TMC12/PR24
Statistical Analysis 3: Comparison: TMC24/PR24 50 mg vs PR48 Control; The difference in the percentage of participants between The TMC24/PR24 50 mg treatment group and the PR48 control group; Test type: Superiority or Other; Difference in percentage of participants = -23.3, 95% CI 2-sided [-59.9 to 19.4] — PR48 control minus TMC24/PR24
Statistical Analysis 4: Comparison: TMC24/PR24 100 mg vs PR48 Control; The difference in the percentage of participants between The TMC24/PR24 100 mg treatment group and the PR48 control group; Test type: Superiority or Other; Difference in percentage of participants = -32.3, 95% CI 2-sided [-66.6 to 8.3] — PR48 control minus TMC24/PR24

7. Primary Outcome: Actual Plasma Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Values up to Week 24 in the Post-treatment Follow-up Period
Description: The table below shows the mean (standard deviation) of the actual HCV RNA values by treatment group at Baseline and Weeks 4, 12, 24, 48, end of treatment (EOT, up to Weeks 24 or 48), Weeks 60 and 72 (Week 24 in the post-treatment follow-up period). The number of participants analyzed is listed at each time point in order of the treatment groups from left to right in the table (ie, Week x, n=x, x, x, x, and x) if different from the "Number of Participants Analyzed." NOTE: All outcome measures reported in this study are "Exploratory;" not "Primary" as indicated (refer to Limits and Caveats).
Time Frame: Baseline, Week 4, 12, 24, 48, EOT (up to Week 24 or 48), and Weeks 60 and 72
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | TMC12/PR24 50 mg | TMC12/PR24 100 mg | TMC24/PR24 50 mg | TMC24/PR24 100 mg | PR48 Control
Number analyzed (Participants) | 27 | 27 | 13 | 13 | 11
log10 IU/mL
  Baseline | 6.19 (0.61) | 6.16 (0.48) | 6.16 (0.44) | 6.43 (0.42) | 6.10 (0.38)
  Week 4 (n=27, 24, 12, 13, and 11) | 0.98 (0.05) | 0.95 (0.0) | 0.98 (0.06) | 0.97 (0.04) | 3.38 (1.82)
  Week 12 (n=27, 22, 12, 13, and 11) | 0.95 (0.0) | 0.95 (0.0) | 0.95 (0.0) | 0.95 (0.0) | 1.84 (1.42)
  Week 24 (n=26, 21, 11, 13, and 11) | 1.12 (0.85) | 0.95 (0.0) | 0.95 (0.0) | 0.95 (0.0) | 1.42 (1.16)
  Week 48 (n=25, 20, 12, 13, and 10) | 1.97 (2.08) | 1.22 (1.20) | 1.42 (1.3) | 1.29 (1.21) | 1.11 (0.49)
  Week 60 (n=0, 0, 0 ,0, and 9) | NA (NA) — no participants were analyzed for this time point | NA (NA) — no participants were analyzed for this time point | NA (NA) — no participants were analyzed for this time point | NA (NA) — no participants were analyzed for this time point | 2.90 (2.31)
  Week 72 (n=0, 0, 0 ,0, and 8) | NA (NA) — no participants were analyzed for this time point | NA (NA) — no participants were analyzed for this time point | NA (NA) — no participants were analyzed for this time point | NA (NA) — no participants were analyzed for this time point | 2.70 (1.07)
  EOT (up to Week 24 or 48) | 1.12 (8.4) | 0.95 (0.0) | 1.17 (0.76) | 0.95 (0.0) | 1.28 (1.07)

8. Primary Outcome: The Number of Participants With Alanine Aminotransaminase (ALT) Values Within the Normal Range at the End-of-treatment (EOT)
Description: The table below shows the number of participants whose ALT results were within the normal range on Day 1 (initial day of treatment), Week 24, 48, and EOT (up to Weeks 24 or 48).The number of participants analyzed is listed at each time point in order of the treatment groups from left to right in the table (ie, Week x, n=x, x, x, x, and x) if different from the "Number of Participants Analyzed." NOTE: All outcome measures reported in this study are "Exploratory;" not "Primary" as indicated (refer to Limits and Caveats).
Time Frame: Day 1, Weeks 24, 48, and EOT (up to Weeks 24 or 48)
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- All TMC435: TMC435 50 mg or 100 mg capsule orally once daily for 12 or 24 weeks
Arm/Group | TMC12/PR24 50 mg | TMC12/PR24 100 mg | TMC24/PR24 50 mg | TMC24/PR24 100 mg | All TMC435 | PR48 Control
Number analyzed (Participants) | 27 | 24 | 13 | 13 | 77 | 11
Participants
  Day 1 (n=27, 24, 13, 13, 77, and 11) | 15 | 15 | 7 | 7 | 44 | 7
  Week 24 (n=26, 21, 11, 13, 71, and 11) | 24 | 18 | 11 | 11 | 64 | 8
  Week 48 (n=25, 20, 12, 13, 70, and 10) | 24 | 20 | 12 | 12 | 68 | 8
  EOT (Weeks 24 or 48) | 23 | 24 | 13 | 11 | 71 | 9

9. Primary Outcome: The Percentage of Participants With Sustained Virologic Response (SVR)
Description: The table below shows the percentage of participants with a SVR4, SVR12, and SVR24 defined as undetectable plasma hepatitis C virus (HCV) ribonucleic acid (RNA) at the end of treatment (EOT) (up to Weeks 24 or 48) and at 4, 12, and 24 weeks, respectively, after the last dose of treatment. NOTE: All outcome measures reported in this study are "Exploratory;" not "Primary" as indicated (refer to Limits and Caveats).
Time Frame: SVR4 (up to Week 28 or Week 52), SVR12 (up to Weeks 36 or 60), and SVR24 (up to Weeks 48 or 72)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC12/PR24 50 mg | TMC12/PR24 100 mg | TMC24/PR24 50 mg | TMC24/PR24 100 mg | PR48 Control
Number analyzed (Participants) | 27 | 24 | 13 | 13 | 11
Percentage of participants
  SVR4 (up to Week 28 or 52) | 88.9 | 95.8 | 92.3 | 92.3 | 63.6
  SVR12 (up to Week 36 or 60) | 85.2 | 79.2 | 84.6 | 92.3 | 45.5
  SVR24 (up to Week 48 or 72) | 77.8 | 79.2 | 76.9 | 92.3 | 45.5

10. Primary Outcome: Predose Plasma Concentrations (C0h) of TMC435 (Sparse Blood Sampling)
Description: The table below shows the mean (standard deviation) predose plasma concentration (C0h) for participants in each treatment group at Weeks 4, 12, and 24. The number of participants analyzed is listed at each time point in order of the treatment groups from left to right in the table (ie, Week x, n=x, x, x, x, and x) if different from the "Number of Participants Analyzed." NOTE: All outcome measures reported in this study are "Exploratory;" not "Primary" as indicated (refer to Limits and Caveats).
Time Frame: Weeks 4, 12, and 24
Population: Pharmacokinetic (PK) analysis was performed in the PK population defined as all participants from whom sparse blood samples were drawn and who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TMC12/PR24 50 mg | TMC12/PR24 100 mg | TMC24/PR24 50 mg | TMC24/PR24 100 mg
Number analyzed (Participants) | 20 | 22 | 10 | 9
ng/mL
  Week 4 (n=20, 22, 10, and 9) | 238 (207) | 1229 (1573) | 194 (156) | 1816 (1429)
  Week 12 (n=26, 20, 12, and 12) | 261 (237) | 1483 (1825) | 221 (209) | 2546 (3011)
  Week 24 (n=0, 0, 10, 10) | NA (NA) — There were no samples for analysis at Week 24. | NA (NA) — There were no samples for analysis at Week 24. | 310 (322) | 2204 (3002)

11. Primary Outcome: Predose Plasma Concentrations (C0h) of TMC435 (Intensive Blood Sampling)
Description: The table below shows the mean predose plasma concentration (C0h) for participants in the 2 TMC435 50 mg treatment groups combined and for participants in the 2 TMC435 100 mg treatment groups combined who had intensive blood samples collected at Weeks 4 to 6. NOTE: All outcome measures reported in this study are "Exploratory;" not "Primary" as indicated (refer to Limits and Caveats).
Time Frame: Weeks 4 to 6
Population: Pharmacokinetic (PK) analysis was performed in the PK population defined as all participants from whom intensive blood samples were drawn and who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TMC435 50 mg | TMC435 100 mg
Number analyzed (Participants) | 14 | 12
ng/mL | 192 (134) | 1732 (2669)

12. Primary Outcome: The Area Under the Plasma Concentration-time Curve From the Time of Administration up to 24 Hours After Dosing (AUC24) for TMC435
Description: The table below shows the mean AUC24 of TMC435 for participants in the 2 TMC435 50 mg treatment groups combined (TMC12/PR24 50 mg and TMC24/PR24 50 mg) and for participants in the 2 TMC435 100 mg treatment groups combined (TMC12/PR24 100 mg and TMC24/PR24 100 mg) who had intensive blood samples collected at Weeks 4 to 6. NOTE: All outcome measures reported in this study are "Exploratory;" not "Primary" as indicated (refer to Limits and Caveats).
Time Frame: within 15 minutes and at 1, 2, 4, 6, 8, 12, and 24 hours post-dose between Week 4 and Week 6 after the initiation of treatment
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ng∙h/mL
Arm/Group | TMC435 50 mg | TMC435 100 mg
Number analyzed (Participants) | 14 | 12
ng∙h/mL | 11182 (7763) [3.95 to 8.00] | 60197 (65364) [4.00 to 12.0]

13. Primary Outcome: Time to Reach the Maximum Plasma Concentration (Tmax) of TMC435
Description: The table below shows the median time in hours to reach the maximum plasma concentration (tmax) of TMC435 for participants in the 2 TMC435 50 mg treatment groups combined (TMC12/PR24 50 mg and TMC24/PR24 50 mg) and for participants in the 2 TMC435 100 mg treatment groups combined (TMC12/PR24 100 mg and TMC24/PR24 100 mg) who had intensive blood samples collected at Weeks 4 to 6. NOTE: All outcome measures reported in this study are "Exploratory;" not "Primary" as indicated (refer to Limits and Caveats).
Time Frame: as for outcome 12
Population: as for outcome 11
Measure: Median (Full Range); unit: Hours
Arm/Group | TMC435 50 mg | TMC435 100 mg
Number analyzed (Participants) | 14 | 12
Hours | 5.97 (725) [3.95 to 8.00] | 6.00 (3446) [4.00 to 12.0]

14. Primary Outcome: The Number of Participants Who Met Virologic Stopping/Continuation Rules and Completed All Study Medications
Description: The table below shows the number of participants who met response-guided treatment (RGT) stopping criteria in the TMC435 treatment groups. Participants who achieved plasma hepatitis C virus (HCV) ribonucleic acid (RNA) levels less than 1.4 log10 IU/mL at Week 4 and had undetectable plasma HCV RNA at Weeks 12, 16 and 20 were to stop all study medication (TMC435, PegIFNα-2a, and ribavirin) at Week 24. All other participants continued PegIFNα-2a and ribavirin until Week 48. NOTE: All outcome measures reported in this study are "Exploratory;" not "Primary" as indicated (refer to Limits and Caveats).
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | TMC12/PR24 50 mg | TMC12/PR24 100 mg | TMC24/PR24 50 mg | TMC24/PR24 100 mg | PR48 Control
Number analyzed (Participants) | 27 | 26 | 13 | 13 | 11
Participants | 25 | 22 | 10 | 12 | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 52 weeks (includes all serious and other adverse events that newly occurred or worsened after treatment with TMC435, PegIFNα-2b or ribavirin, until the end date of the last study medication intake + 28 days).
Arm/Group | TMC12/PR24 50 mg | TMC12/PR24 100 mg | TMC24/PR24 50 mg | TMC24/PR24 100 mg | PR48 Control
Serious Adverse Events (participants affected / at risk) | 0/27 | 3/26 | 1/13 | 1/13 | 0/13
Other Adverse Events (participants affected / at risk) | 27/27 | 26/26 | 13/13 | 13/13 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TMC12/PR24 50 mg (N=27) | TMC12/PR24 100 mg (N=26) | TMC24/PR24 50 mg (N=13) | TMC24/PR24 100 mg (N=13) | PR48 Control (N=13)
Malaise (General disorders) | 0 | 1 | 0 | 0 | 0
Incorrect dose administered (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Vulvar erosion (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TMC12/PR24 50 mg (N=27) | TMC12/PR24 100 mg (N=26) | TMC24/PR24 50 mg (N=13) | TMC24/PR24 100 mg (N=13) | PR48 Control (N=13)
Anaemia (Blood and lymphatic system disorders) | 8 | 6 | 5 | 5 | 5
Palpitations (Cardiac disorders) | 1 | 1 | 0 | 0 | 2
Dermoid cyst (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 0 | 2 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Thyroid disorder (Endocrine disorders) | 0 | 0 | 0 | 1 | 0
Asthenopia (Eye disorders) | 1 | 0 | 1 | 1 | 1
Cataract (Eye disorders) | 0 | 0 | 0 | 1 | 0
Conjunctival deposit (Eye disorders) | 0 | 0 | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 1 | 1 | 0 | 0
Keratoconjunctivitis sicca (Eye disorders) | 0 | 0 | 0 | 0 | 1
Macular oedema (Eye disorders) | 0 | 0 | 0 | 1 | 0
Ocular discomfort (Eye disorders) | 0 | 0 | 1 | 0 | 0
Punctate keratitis (Eye disorders) | 0 | 0 | 1 | 0 | 0
Retinal degeneration (Eye disorders) | 0 | 0 | 0 | 0 | 1
Retinal exudates (Eye disorders) | 1 | 2 | 1 | 2 | 0
Retinal haemorrhage (Eye disorders) | 0 | 2 | 1 | 0 | 1
Retinal vein occlusion (Eye disorders) | 1 | 0 | 0 | 1 | 0
Retinopathy (Eye disorders) | 0 | 2 | 0 | 1 | 3
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 1
Vitreous floaters (Eye disorders) | 0 | 0 | 1 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 6 | 3 | 3 | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 4 | 1 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 4 | 1 | 1 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 4 | 6 | 3 | 0 | 5
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Faeces hard (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 5 | 5 | 2 | 1 | 0
Periodontitis (Gastrointestinal disorders) | 1 | 3 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 7 | 5 | 5 | 2 | 2
Tongue disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2 | 2 | 2
Chest discomfort (General disorders) | 0 | 0 | 2 | 0 | 0
Chills (General disorders) | 1 | 1 | 1 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 2 | 0 | 0
Feeling abnormal (General disorders) | 0 | 0 | 1 | 0 | 1
Feeling cold (General disorders) | 0 | 0 | 0 | 1 | 1
Injection site erythema (General disorders) | 3 | 2 | 1 | 2 | 1
Injection site pruritus (General disorders) | 1 | 1 | 0 | 0 | 1
Injection site reaction (General disorders) | 7 | 2 | 6 | 5 | 3
Malaise (General disorders) | 17 | 15 | 8 | 7 | 8
Pyrexia (General disorders) | 18 | 10 | 7 | 7 | 7
Thirst (General disorders) | 0 | 1 | 1 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 5 | 2 | 3 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 2 | 0 | 0 | 1 | 1
Enteritis infectious (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 9 | 4 | 4 | 2 | 3
Onychomycosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Oral herpes (Infections and infestations) | 1 | 2 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 3 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0 | 1 | 1
Alpha-1 acid glycoprotein increased (Investigations) | 5 | 1 | 2 | 0 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 1 | 1
Blood amylase increased (Investigations) | 0 | 0 | 0 | 2 | 0
Blood bilirubin increased (Investigations) | 3 | 6 | 1 | 3 | 0
Blood calcium decreased (Investigations) | 1 | 0 | 2 | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 2 | 2 | 0 | 2
Blood phosphorus decreased (Investigations) | 2 | 0 | 1 | 2 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 1 | 1 | 1
Blood triglycerides increased (Investigations) | 1 | 1 | 2 | 2 | 3
Blood uric acid increased (Investigations) | 4 | 2 | 1 | 0 | 0
Electrocardiogram T wave inversion (Investigations) | 0 | 0 | 1 | 0 | 0
Haematocrit decreased (Investigations) | 4 | 6 | 4 | 3 | 4
Haemoglobin decreased (Investigations) | 8 | 12 | 7 | 7 | 6
Lipase increased (Investigations) | 0 | 2 | 0 | 3 | 1
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 1 | 0
Mean cell haemoglobin concentration decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Mean cell volume increased (Investigations) | 0 | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 12 | 14 | 10 | 12 | 9
Platelet count decreased (Investigations) | 5 | 4 | 4 | 6 | 6
Protein urine present (Investigations) | 0 | 0 | 1 | 0 | 2
Red blood cell count decreased (Investigations) | 4 | 6 | 5 | 3 | 4
Tri-iodothyronine free decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 1 | 3 | 2 | 0 | 2
White blood cell count decreased (Investigations) | 16 | 15 | 10 | 12 | 10
White blood cells urine positive (Investigations) | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 4 | 6 | 4 | 1 | 3
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1
Hypo HDL cholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypocholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 7 | 6 | 5 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 1 | 2 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 6 | 4 | 1 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 1 | 0 | 0
Dizziness postural (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 3 | 1 | 1 | 1 | 0
Head discomfort (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 14 | 13 | 8 | 6 | 8
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 2 | 1 | 0 | 1 | 0
Syncope (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Anxiety disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0
Depressive symptom (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 10 | 5 | 5 | 3 | 2
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Cystitis-like symptom (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1
Galactorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 0 | 1 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 0 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 11 | 6 | 5 | 3 | 6
Asteatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 2 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 4 | 0 | 6 | 0
Rash (Skin and subcutaneous tissue disorders) | 17 | 15 | 7 | 8 | 6
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 4 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 3 | 0 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
All outcome measures reported in this study are "Exploratory;" not "Primary" as indicated. "Primary" was chosen for each outcome measure because "Exploratory" is not available as an outcome measure type.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.